CLINICAL TRIAL: NCT07344415
Title: Level of Anxiety During Caries Removal Using a New Chemo-mechanical Caries Removal System Versus Conventional Drilling Method: A Randomized Controlled Trial
Brief Title: Anxiety During Caries Removal Using Chemo-mechanical Versus Conventional Methods
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmine Ashraf Elbanna, Lecturer, Department of Conservative Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cariemove
Record Dates: First submitted 2025-12-28; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Caries Active
Keywords: Chemo-mechanical; Rotary; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemo-mechanical (Experimental)
  Interventions: Procedure: Cariemove
- Conventional rotary (Active Comparator)
  Interventions: Procedure: Drilling using bur

INTERVENTIONS:
Procedure: Cariemove — It is a newly introduced Egyptian product. It consists of a transparent liquid containing 0.5% sodium hypochlorite, 0.1 M mixtures of three amino acids, leucine, lysine and glutamic acid.
  Arms: Chemo-mechanical
Procedure: Drilling using bur — Rotary dental burs using high speed hand piece under water spray cooling system
  Arms: Conventional rotary

SUMMARY:
This study aims to clinically assess this newly introduced Egyptian chemo-mechanical caries removal gel versus conventional drilling method . The concept of preserving healthy tooth structures and employing atraumatic restorative techniques during cavity preparation aligns with the principles of minimally invasive dentistry. This approach prioritizes patient comfort, reassurance, and fosters a positive perception of dental treatment.

DETAILED DESCRIPTION:
Dental caries is a multifactorial dynamic disease that involves mineral loss of dental hard tissue. Caries management is the action made to interfere with the loss of minerals that could be non-operative or operative interventions according to the stage and severity of the case. In deep carious lesions, removal of caries using rotary instruments has been the most prevalent technique. This could be attributed to being rapid and efficient in caries removal. However, such technique possesses some drawbacks in terms of patient discomfort, thermal stimulation to the pulp and unnecessary excessive removal of tissues. Minimally invasive dentistry is the philosophy that aims for lesion control as well as minimal operative intervention. Preserving dental tissue by early caries detection of as well as combining non-operative minimally invasive restorative procedures are its main objective. Therefore, alternative techniques have been proposed to overcome the drawbacks of rotary instrumentation of deep lesions. One of the techniques is chemico-mechanical caries removal. Chemico-mechanical caries removal is based on enzymatic action on carious tissues dissolving them to be easily removed using an excavator. Such system allows better patient perception by avoiding the vibration caused by rotary instruments. It also helps in avoiding excessive pulpal irritation caused by the heat generated while using rotary instruments. Cariemove ,a newly introduced Egyptian product, that is based on amino acids, sodium hypochlorite and carboxyglyciene has been introduced in the market. This system lacks sufficient literature about its clinical efficiency and level of anxiety of patients during caries removal.

ELIGIBILITY:
Inclusion Criteria:

1. Open carious lesions with dentin involvement, but not involving the pulp in lower molars.
2. The access of the carious lesion has to be large enough to allow the penetration of the excavator.
3. Asymptomatic vital teeth, without clinical evidence of pulp, furcation, or periapical pathology.
4. Patients who sign informed consent.
5. Co-operative patients approving to participate in the trial.

Exclusion Criteria:

1. Patients with spontaneous or elicited pain from caries.
2. Patients with systemic diseases.
3. Presence of intraoral/extraoral swellings.
4. Deep dental caries involving pulp.
5. Presence of swelling/fistula in relation to carious tooth.
6. Inability to return for recall visits.
7. Patients with bad oral hygiene
8. Refuse to participate in the study.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Level of anxiety and discomfort | Baseline (Day 1)
  Visual Analogue Scale from 0 to 10 (0 represents no pain and 10 represents the worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of privacy concerns and institutional policy restrictions.